CLINICAL TRIAL: NCT04747405
Title: Evaluation of Psychological Impact of Group Therapy for Patients Who Have Been Hospitalized in Intensive Care During COVID-19 Pandemic: Exploratory Study
Acronym: GPR COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHMS20009
Record Dates: First submitted 2021-02-09; First posted 2021-02-10 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Intensive Care Unit Syndrome; Covid19; Anxiety; Depression
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Depression | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A standard (No Intervention): standard of care
- B therapy group (Experimental): standard of care and therapy group
  Interventions: Other: therapy group

INTERVENTIONS:
Other: therapy group — therapy group of maximum 8 people repeated twice
  Arms: B therapy group

SUMMARY:
Psychological impact of intensive care hospitalization for patients has been demonstrated during the last few years: anxiety, depression and post traumatic stress disorder. Hospitalizations during COVID-19 pandemic have been marked by factors such as confinement forbidding family members visits, stress on intensive care unit ...Those factors may have a psychological impact added to factors of long hospitalization and prolonged mechanical ventilation.

For all these reasons the investigators fear that patients hospitalized in intensive care during COVID-19 pandemic develop psychological trouble with an increased risk for those who experienced COVID-19 infection. The hypothesis therapy group added to standard care might have a positive impact on psychological troubles such as anxiety, depression and post traumatic stress disorder for patients who have been hospitalized in intensive care during COVID-19 pandemic.

The investigators will compare two groups:

* group receiving standard of care
* group receiving standard of care and therapy group

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* hospitalized at least 72h in intensive care during COVID-19 pandemic crisis
* out of intensive care for at least 2 months and maximum 6 months
* psychological evaluation done according to local practice and standard of care
* speaking french
* patient coming alone to the therapy group
* patient agree to respect confidentiality rules and demonstrating goodwill with others participants
* patient comite to respecting barriers rules against COVID-19
* affiliated to social security system
* no juridic protection engaged

Exclusion Criteria:

* presenting psychological disease
* drug addiction
* participation to other interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
prevalence of post traumatic stress syndrome | 12 months after intensive care hospitalization
  the aim is to compare the prevalence of post traumatic stress syndrome between both groups 12 months after exiting intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Romain PERCOT, Study Director — Cebtre Hospitalier Metropole Savoie
Locations (1):
- CH Métropole Savoie, Chambéry, France

IPD SHARING:
Plan to Share IPD: No